CLINICAL TRIAL: NCT03421028
Title: The Evaluation of EMG-biofeedback Therapy Efficiency in Management of Masticatory Muscles Pain
Brief Title: Evaluation of Biofeedback Therapy Efficiency in Masticatory Muscles Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Wojciech Florjański, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMU2/2017
Record Dates: First submitted 2018-01-02; First posted 2018-02-05 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Muscle Pain; Feedback, Psychological; Craniomandibular Disorders; Temporomandibular Disorder; Sleep
MeSH Terms: conditions — Myalgia; Craniomandibular Disorders; Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Patients with masticatory muscle pain treated with occlusal splint, physiotherapy and counseling
  Interventions: Other: Classic treatment for myogenous TMD
- Experimental group 1 (Experimental): Patients diagnosed with masticatory muscle pain treated with 4 meetings of EMG-biofeedback assisted training
  Interventions: Device: Electromyography Biofeedback
- Experimental group 2 (Experimental): Patients diagnosed with masticatory muscle pain treated with 8 meetings of EMG-biofeedback
  Interventions: Device: Electromyography Biofeedback

INTERVENTIONS:
Device: Electromyography Biofeedback — EMG-Biofeedback- assisted training is a method in which electrodes situated on the surface of the skin detect small voltage changes which arise from the working muscles (in this case masseter and temporalis muscles). The voltage is transformed into a visual or sound time-variable signal which gives the patient feedback as he willingly tries to change the muscle tension (in this case to lower the excessive masseter tension)
  Other Names: EMG-Biofeedback
  Arms: Experimental group 1; Experimental group 2
Other: Classic treatment for myogenous TMD — Combination of physiotherapy (manual therapy), stabilization occlusal splint usage and counseling
  Arms: Control group

SUMMARY:
This study evaluates beneficial effects of biofeedback therapy in reducing pain and increased tension of muscles occurring in patients with temporomandibular disorders (TMD). During the study Electromyography Biofeedback (EMG-Biofeedback)- assisted training lowering muscle tension will be used. The patients will undergo 4 or 8 meetings of EMG-Biofeedback - assisted training Than the patients will be reevaluated after 6 and 12 weeks.

DETAILED DESCRIPTION:
1. The Aim:

   The aim of the study is to evaluate beneficial effects of biofeedback therapy in reducing pain, increased tension of masticatory muscles occurring in patients with myogenous TMD and if the therapy influences psychological and sleep parameters. Also to verify if the effect of the therapy persists in time.
2. Patients:

   1. Experimental group 1 - patients diagnosed with myalgia subjected to 4 EMG-Biofeedback trainings. The group will include approximately 20 adults.
   2. Experimental group 2 - patients diagnosed with myalgia subjected to 8 EMG-Biofeedback trainings. The group will include approximately 20 adults.
   3. Control group - patients diagnosed with myalgia subjected to physiotherapy (manual therapy), stabilization splint usage and counseling (20 adults).
3. Methods:

Adult patients diagnosed with masticatory muscles myalgia will be included in this study. All participants will be evaluated in accordance to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD). Intensity of pain in the masticatory muscles will be defined using the Numerical Rating Scale (NRS). The pressure pain threshold (PPT) will be assessed with an dolorimeter and noticed on DC/TMD pain drawing diagram. Each of the qualified patients will also undergo the electromyography of temporal and masseter muscles. All participants will fill in questionnaires (Graded Chronic Pain Scale (GCPS), Pittsburgh Sleep Quality Index (PSQI), Patient Health Questionnaire-9 (PHQ-9), Beck Anxiety Inventory (BAI) and Perceived Stress Scale-10 (PSS-10) and Somatic Symptom Scale-8 (SSS-8).

Patients qualified to the experimental groups will be divided in to 2 subgroups composed of 20 participants each.

Experimental group 1 will undergo a cycle of 4 meetings (1 per week) of 20 minute EMG-Biofeedback- assisted training decreasing the masseter and temporalis muscle tension. 10 minutes of training for each group of muscle.

Experimental group 2 will undergo a cycle of 8 meetings (1 per week) of 20 minute EMG-Biofeedback- assisted training decreasing the masseter and temporalis muscle tension. 10 minutes of training for each group of muscle.

Postcycle examination:

After completing the cycle, patients from the study group and control group will be reevaluated. All participants will be evaluated in accordance to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD). Intensity of pain in the masticatory muscles will be defined using the Numerical Rating Scale (NRS). The pressure pain threshold (PPT) will be assessed with an dolorimeter and noticed on DC/TMD pain drawing diagram. Each of the qualified patients will also undergo the electromyography of temporal and masseter muscles. All participants will fill in questionnaires (Graded Chronic Pain Scale (GCPS), Pittsburgh Sleep Quality Index (PSQI), Patient Health Questionnaire-9 (PHQ-9), Beck Anxiety Inventory (BAI) and Perceived Stress Scale-10 (PSS-10) and Somatic Symptom Scale-8 (SSS-8).

The postcycle examination will take place after last planned training and during follow-ups - 6 and 12 weeks after completion of EMG-Biofeedback therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of myalgia in accordance to Diagnostic Criteria for Temporomandibular Disorders
* full dentition or single tooth loss
* age between 18 and 70

Exclusion Criteria:

* age under 18
* age over 70
* terminal general diseases
* severe mental disorders
* severe neurological disorders
* intake of drugs affecting muscle function
* edentulism or destruction of dentition
* alcoholism
* drug addiction
* history of severe trauma in the head and neck region
* severe pathology of temporomandibular joints
* congenital or acquired craniofacial deformity
* patients suffering from neuropathic pain
* patients with craniofacial inflammation
* patients undergoing orthodontic treatment
* pregnancy
* significant postural defect

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of EMG biofeedback therapy on pain symptoms measured by Numerical Rating Scale (NRS) in Experimental group 1 | before the treatment, after 4 weeks of training
  This effect will be assessed by comparing Numerical Rating Scale (NRS) pre- and post- biofeedback therapy. A numerical rating scale (NRS) requires the patient to rate their pain on a scale 0-10, where 0 is no pain and 10 is the worst pain imaginable
The effect of EMG biofeedback therapy on pain symptoms measured by Numerical Rating Scale (NRS) in Experimental group 2 | before the treatment, after 8 weeks of training
  This effect will be assessed by comparing Numerical Rating Scale (NRS) pre- and post- biofeedback therapy. A numerical rating scale (NRS) requires the patient to rate their pain on a scale 0-10, where 0 is no pain and 10 is the worst pain imaginable
The effect of EMG biofeedback therapy on pain symptoms measured by pressure pain threshold in Experimental group 1 | before the treatment, after 4 weeks of training
  This effect will be assessed by comparing pressure pain threshold pre- and post- biofeedback therapy. Pressure pain threshold will be measured with dolorimeter.
The effect of EMG biofeedback therapy on pain symptoms measured by pressure pain threshold in Experimental group 2 | before the treatment, after 8 weeks of training
  This effect will be assessed by comparing pressure pain threshold pre- and post- biofeedback therapy. Pressure pain threshold will be measured with dolorimeter.

SECONDARY OUTCOMES:
Effect of EMG biofeedback therapy on psychological parameters and its persistence in time measured by Beck Anxiety Inventory (BAI). | before the treatment and up to 12 weeks after completion of the treatment
  This effect will be assessed by comparing the results of Beck Anxiety Inventory. Each participant will fill in Beck Anxiety Inventory pre- post therapy and during the follow-ups. The total score is calculated by finding the sum of the 21 items. Total score for all 21 symptoms that can range between 0 and 63 points. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and; 26 - 63 as "Severe".
Effect of EMG biofeedback therapy on psychological parameters and its persistence in time measured by Patient Health Questionnaire-9 (PHQ-9) | before the treatment and up to 12 weeks after completion of the treatment
  This effect will be assessed by comparing the results of Patient Health Questionnaire-9 (PHQ-9) . Each participant will fill in Patient Health Questionnaire - 9 pre- post therapy and during the follow-ups. PHQ-9 total score for the nine items ranges from 0 to 27.Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Effect of EMG biofeedback therapy on psychological parameters and its persistence in time measured by Perceived Stress Scale-10 (PSS-10) | before the treatment and up to 12 weeks after completion of the treatment
  This effect will be assessed by comparing the results of Perceived Stress Scale-10 (PSS-10). Each participant will fill in Perceived Stress Scale -10 pre- post therapy and during the follow-ups. Scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. It can range from 0 to 40. Scores ranging from 0-13 would be considered low stress,14-26 would be considered moderate stress, 27-40 would be considered high perceived stress.
Effect of EMG biofeedback therapy on psychological parameters and its persistence in time measured by Somatic Symptom Scale-8 (SSS-8). | before the treatment and up to 12 weeks after completion of the treatment
  This effect will be assessed by comparing the results Somatic Symptom Scale-8 (SSS-8). Each participant will fill in Somatic Symptom Scale-8 (SSS-8) pre- post therapy and during the follow-ups. SSS-8 total score ranges from 0 to 32 points, where 0-3 points means no to minimal severity, 4-7 points - low severity, 8-11 points - medium severity, 12-15 points - high severity, 16-32 points - very high severity.
Effect of EMG biofeedback therapy on sleep quality and its persistence in time measured by Pittsburgh Sleep Quality Index (PSQI) | before the treatment and up to 12 weeks after completion of the treatment
  This effect will be assessed by comparing the results of Pittsburgh Sleep Quality Index (PSQI). Each participant will fill in Pittsburgh Sleep Quality Index pre- post therapy and during the follow-ups. The measure consists of 19 individual items, creating 7 components that produce one global score ranging from 0 to 21, where lower scores mean better sleep quality.
Effectiveness of EMG biofeedback therapy on pain symptoms in comparison to "standard" treatment measured by Numerical Rating Scale (NRS) | after treatment and up to 12 weeks later
  This effect will be assessed by comparing Numerical Rating Scale (NRS) between studied and control group. The results will be compared after treatment and during follow-ups. A numerical rating scale (NRS) requires the patient to rate their pain on a scale 0-10, where 0 is no pain and 10 is the worst pain imaginable
Effectiveness of EMG biofeedback therapy on pain symptoms in comparison to "standard" treatment measured by pressure pain threshold | after treatment and up to 12 weeks later
  This effect will be assessed by comparing pressure pain threshold measured with dolorimeter between studied and control group. The results will be compared after treatment and during follow-ups.
Persistence in time of EMG biofeedback therapy effects on pain symptoms measured by Numerical Rating Scale (NRS) | after treatment and up to 12 weeks later
  This effect will be assessed by comparing Numerical Rating Scale (NRS) pre- and post- biofeedback therapy. A numerical rating scale (NRS) requires the patient to rate their pain on a scale 0-10, where 0 is no pain and 10 is the worst pain imaginable
Persistence in time of EMG biofeedback therapy effects on pain symptoms measured by pressure pain threshold | after treatment and up to 12 weeks later
  This effect will be assessed by comparing pressure pain threshold pre- and post- biofeedback therapy. Pressure pain threshold will be measured with dolorimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Mieszko Więckiewicz, D.M.D.Ph.D., Study Chair — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Dolny Śląsk, Poland

IPD SHARING:
Plan to Share IPD: No